CLINICAL TRIAL: NCT06630169
Title: APANECA: A Prospective, Parallel-arm, Multi-Surgeon Study of Cryopreserved AURN001 in Subjects With Corneal Edema Secondary to Corneal Endothelial Dysfunction (2024-E002-C)
Brief Title: Study of Cryopreserved AURN001 in Subjects With Corneal Edema Secondary to Corneal Endothelial Dysfunction
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aurion Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APANECA
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Corneal Edema
MeSH Terms: conditions — Corneal Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Other): Endothelial polishing zone 1 (low)
  Interventions: Combination Product: Cryopreserved AURN001
- Arm 2 (Other): Endothelial polishing zone 2 (medium)
  Interventions: Combination Product: Cryopreserved AURN001
- Arm 3 (Other): Endothelial polishing zone 3 (high)
  Interventions: Combination Product: Cryopreserved AURN001

INTERVENTIONS:
Combination Product: Cryopreserved AURN001 — Corneal Endothelial Cells and Y27632

SUMMARY:
The purpose of this study is to assess the safety and efficacy of cryopreserved AURN001 in patients with corneal edema secondary to endothelial dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of corneal edema secondary to corneal endothelial dysfunction, requiring surgery (full- or partial-thickness endothelial keratoplasty)
* BCVA no worse than 5 ETDRS letters (i.e., 1.6 LogMAR or approximate 20/800 Snellen equivalent).

Exclusion Criteria:

* Have pre-operative corneal epithelial, sub-epithelial or stromal scarring or other opacity that is paracentral/central and visually significant, but not suspected to be secondary to corneal endothelial disease with the potential to improve from treatment in the study eye
* Have history or presence of an ocular disease other than corneal endothelial dysfunction that could affect vision or safety assessments

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-09-16 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
BCVA - 15-letter improvement (3-line gain) | Month 6
  Response, defined as a ≥15-letter improvement (3-line gain) from baseline in best-corrected visual acuity (BCVA)

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, OD, Study Director — Aurion Biotech
Locations (1):
- Aurion Biotech site, San Salvador, El Salvador